CLINICAL TRIAL: NCT05975242
Title: Acceptability and Impact of the Proactive Use of a Diabetes Management Smartphone Application (mySugr) for Spanish-literate Adults With Poorly Controlled Non-intensively Treated Type 2 Diabetes
Brief Title: Acceptability & Impact of a Diabetes Management Smartphone App (mySugr) for Spanish-literate Adults With Type 2 Diabetes
Acronym: mySugr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIS-000011
Record Dates: First submitted 2023-07-27; First posted 2023-08-03 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Hispanic/Latino; smartphone application; self-monitoring blood glucose; Spanish; mySugr PRO
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study will be single site, prospective data collection, with pre- and post-intervention comparison. A total of 30 people with T2D will be randomly allocated (2:1 randomization) to the interventional group (n = 20) that will use the digital self-management application during the 12-week study period or the control group (n = 10) without the app.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): The interventional group will use the digital self-management smartphone application during the 12-week study period and will have access to 3 coaching sessions. The interventional group will be trained in the use of the app and receive education focused on self-monitoring blood glucose based on paired (before and 2 hours after a meal) blood glucose testing, which participants will conduct twice daily for 6 days once monthly for 3 months.
  Interventions: Behavioral: Smartphone diabetes management application
- Control group (No Intervention): The control group will not have use of the digital self-management smartphone application during the 12-week study period and will not have access to 3 coaching sessions. No structured self-monitoring blood glucose testing will be done.

INTERVENTIONS:
Behavioral: Smartphone diabetes management application — The intervention is a smartphone diabetes management application that is combined with structured blood glucose testing.
  Other Names: mySugr
  Arms: Interventional group

SUMMARY:
The goal of this clinical trial is to compare those using a diabetes management smartphone application (mySugr) to those not using the application. This smartphone application is for Spanish-literate adults with poorly controlled, non-intensively treated type 2 diabetes (T2D).

The main question[s] that it aims to answer are:

* What is the impact of the use of mySugr (a smartphone-based application or app) with structured blood glucose monitoring on diabetes self-management among Hispanic/Latino adults with poorly controlled, non-intensively treated T2D?
* Will diabetes self-management be more effective for those using mySugr (the Active group) compared to those not using mySugr (the Control group) over a 12-week study period? Participants will be screened and enrolled if they are eligible; they will have the study explained to them in Spanish or English and have time to ask questions and then sign an informed consent form. Clinical measurements (including height, weight, and blood pressure) and hemoglobin A1c will be done. All subjects will be given a blood glucose meter, lancing device, and blood glucose strips for the meter, and they will also receive an electronic scale. Several questionnaires will be answered.

If a subject is randomly assigned to the Active group, they will download the mySugr PRO (professional) app in Spanish to their smartphone and be trained in its use. They will receive education focused on paired (before and 2 hours after a meal) blood glucose testing, which participants will conduct twice a day for 6 days and once a month for 3 months. Participants will continue structured blood glucose testing with the mySugr PRO app for 12 weeks, and they will have 3 virtual visits in Spanish with mySugr PRO coaches who will review the blood glucose records and advise the subjects.

Subjects in the Control group will not receive the mySugr PRO app or coaching. They will continue with their usual diabetes management.

All subjects will return after 12 weeks to return the scale and have a close-out visit with clinical measurements and questionnaires. Subjects will also receive a disturbance allowance for their time and participation.

DETAILED DESCRIPTION:
The aim of this pilot observation trial is to determine feasibility, acceptability, and impact of the combination of mySugr and structured self-monitored blood glucose (SMBG) for Spanish-literate Hispanic/Latino adults with poorly controlled T2D. The study will be single site (Sansum Diabetes Research Institute - SDRI), prospective data collection, with pre- and post-intervention comparison. A total of 30 people with T2D will be randomly allocated (2:1 randomization) to the interventional group (n = 20) that will use the digital self-management application during the 12-week study period or the control group (n = 10) without the app. Pre- and post-intervention assessments will measure diabetes distress as well as self-efficacy to manage diabetes, HbA1c, weight, and blood glucose. MySugr app perceived usefulness, ease of use, content, efficacy, and usability will be measured post-intervention. To maximize retention, both participant groups will receive a disturbance allowance as they progress through the study.

Spanish-literate Hispanic/Latino adults with T2D and HbA1c 7.5% - 10% and who reside in the Central Coast of California and currently use a compatible smartphone will be enrolled.

Study interaction and procedures will be conducted in Spanish by an existing, trusted bilingual Hispanic/Latino Certified Diabetes Educator (CDE) and SDRI Community Scientists. Following informed consent, participants will be randomly assigned to the interventional group that will use the digital self-management application during the 12-week study period or the control group that will not use the app. The interventional group will be trained in the use of the mySugr app and receive education focusing on SMBG based on paired (before and 2 hours after a meal) blood glucose (BG) testing, which participants will conduct twice daily for 6 days once monthly for 3 months. Participants will continue structured SMBG with mySugr PRO for 12 weeks and will have access to mySugr proactive coaching consisting of 3 virtual engagements focused on reviewing and reacting to participant-derived structured SMBG data.

At Visit 1, vital signs health measurements (height, weight, waist circumference and resting blood pressure) will be conducted by trained clinical staff, and fingerstick HbA1c will be measured using the Abbott Afinion 2 Point of Care (POC) Analyzer or FDA-approved equivalent. Several questionnaires will be completed. Subjects will measure their blood glucose at home using the Accu Check Guide Me blood glucose meter and their weight at home using a smartphone connected weight scale.

If subjects are randomized to the Active or intervention group, they will download and be trained in the use of the mySugr app. Active group participants will be asked to use the mobile application throughout the duration of the study. The app will be used to collect data from glucometers in their mobile phones and to have access to mySugr proactive coaching. The coach visits will be conducted in Spanish with a duration of 30-minutes each month and focusing on reviewing and reacting to participant derived structured SMBG data. In the control group, people with diabetes will neither have access to the mySugr Pro app nor coaching during the 12-week Intervention Period; they will continue with their usual, discretionary mode of therapy, data documentation, and glucose monitoring.

After 12 weeks, subjects will complete a second and final visit with vital signs, HbA1c, and questionnaires repeated. A disturbance allowance will be given to each subject for their time and participation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age at enrollment
2. Self-reported Hispanic/Latino ethnicity
3. Spanish-literate with Spanish as preferred language
4. Diagnosis of T2D for at least 6 months
5. HbA1c 7.5% - 10%
6. mySugr-compatible smartphone
7. Any glucose lowering therapy except rapid-acting mealtime insulin
8. Residence in Central Coast of California -

Exclusion Criteria:

1. Type 1 diabetes 2. Use of rapid-acting mealtime insulin 3. Pregnancy 4. Any active clinically significant disease or disorder which in the investigator's opinion could interfere with participation in the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Spanish-language Diabetes Self-Efficacy Scale (DSES-S) | Visit 1, week 1 and Visit 2, week 12
  A scale of 8 Likert-type 10-point items to measure self-efficacy of diabetes self-management

SECONDARY OUTCOMES:
Hemoglobin A1c | Visit 1, week 1 and Visit 2, week 12
  A measure of glycosylated hemoglobin
Problem areas in diabetes (PAID) scale | Visit 1, week 1 and Visit 2, week 12
  The Problem Areas in Diabetes (PAID) instrument was developed to measure emotional distress in people with diabetes. It is a 20-item scale consisting of emotional problems commonly reported in type 1 and type 2 diabetes mellitus, and has been found to be a valid and reliable scale in Western populations.
Blood glucose measurements | Week 1, Week 4, Week 8
  Blood glucose measurements made with the assigned glucose meter at specific times
Weight | Visit 1, week 1 and Visit 2, week 12
  Body weight in kilograms

OTHER OUTCOMES:
Health Information Technology Usability Evaluation Scale (Health-ITUES) | Visit 1, week 1 and Visit 2, week 12
  The measurement scale is used to assess perceived usefulness and perceived ease of use.
Mobile App Rating Scale (MARS) | Visit 1, week 1 and Visit 2, week 12
  The measurement scale is used to assess the content, efficacy and usability of a smartphone application.
Mobile Device Proficiency Questionnaire (MDPQ) | Visit 1, week 1 and Visit 2, week 12
  A questionnaire to assess digital literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Thorsell, MD, Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States